CLINICAL TRIAL: NCT07257393
Title: Validation of a Mobile Health Application for Fall Risk Assessment in Parkinson's Disease: A Comparative Study Before and After Dopaminergic Medication Adjustment
Brief Title: Fall Risk Assessment in Parkinson's Disease Using Kinetikos Health
Acronym: PD_FALLRISK
Status: Not yet recruiting | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202511067
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Parkinsonism
Keywords: Parkinson's disease; Fall risk; Motor fluctuation; Dopaminergic medication; Mobile health; Sit-to-Stand; Kinetikos Health App
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opicapone group: PD patients undergo dopaminergic medication adjustments
  Interventions: Other: No Intervention: Observational Cohort
- Safinamide group: PD patients undergoing dopaminergic medication adjustments
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention.

SUMMARY:
This is a single-center, prospective observational study aiming to validate the Kinetikos Health App for fall risk assessment in PD patients undergoing dopaminergic medication adjustments.

DETAILED DESCRIPTION:
Falls are common and disabling in PD. Dopaminergic medication effects on fall risk remain inconclusive. This study validates the Kinetikos Health App for objective fall risk assessment before and after medication adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20;
2. PD diagnosis (MDS criteria);
3. On levodopa monotherapy with motor fluctuations;
4. Planned to start opicapone or safinamide;
5. Consent provided.

Exclusion Criteria:

1. Atypical/secondary parkinsonism;
2. Moderate-severe dementia;
3. DBS/MRgFUS/neurosurgery within 6 months;
4. Severe comorbidities limiting test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from outpatient neurology clinic, Shuang Ho Hospital, Taipei Medical University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in fall-risk index (Kinetikos Health App Sit-to-Stand) | From baseline to 3 months

SECONDARY OUTCOMES:
UPDRS | From baseline to 3 months
  Change in MDS-UPDRS axial score; Change in MDS-UPDRS Part II
Fall events | From baseline to 3 months
  Fall events during 3 months
LEDD | From baseline to 3 months
  Change in LEDD

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Chih Chung, MD, Principal Investigator — Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing; results published in aggregate